CLINICAL TRIAL: NCT00802308
Title: A Randomized, Partially Blind, Four-way Crossover Study to Determine the Effects of a Single Dose of Egalet® Morphine Combined With a Single Dose of Alcohol in Healthy Male and Female Moderate Drinkers
Brief Title: Effects of a Single Dose of Egalet® Morphine Combined With a Single Dose of Alcohol in Healthy Moderate Drinkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: MP-EG-010
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): Single dose administration of Egalet® morphine with alcohol
  Interventions: Drug: Morphine sulphate
- Treatment B (Experimental): Single dose administration of Egalet® morphine with alcohol
  Interventions: Drug: Morphine sulphate
- Treatment C (Experimental): Single dose administration of Egalet® morphine with alcohol
  Interventions: Drug: Morphine sulphate
- Treatment D (Placebo Comparator): Single dose administration of Egalet® morphine with water
  Interventions: Drug: Morphine sulphate

INTERVENTIONS:
Drug: Morphine sulphate — Extended release tablet combined with alcohol or water

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics of Egalet® morphine when administered with alcohol and compare to administration with water.

DETAILED DESCRIPTION:
Outcome: Pharmacokinetic parameters

ELIGIBILITY:
Main Inclusion Criteria:

* Body mass index (BMI) within the range of 20 to 33 kg/m2 and a minimum weight of at least 50 kg.
* Current alcohol users who are classified as moderate drinkers
* Able to abstain from alcohol during the 48 hour period preceding each study visit
* Free from any clinically significant abnormality on the basis of medical history, vital signs, physical examination, 12-Lead ECG, and laboratory evaluation

Main Exclusion Criteria:

* Intolerance towards alcohol
* History of allergy or hypersensitivity to opioids or related drugs or any excipients
* Any history of drug or alcohol dependence
* Clinically significant abnormalities on physical examination, medical history, 12-Lead ECG, vital signs, or laboratory values
* Gastrointestinal disease or constipation or other clinically significant gastrointestinal problems

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To evaluate pharmacokinetic effects of the co-administration of alcohol and Egalet® morphine. AUC0-t, AUC0-inf, Cmax, Residual Area, Tmax, T½ el, and Kel. | Single-dose evaluation

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the co-administration of alcohol and Egalet® morphine. Hematology, biochemistry, urinalysis, ECG, vital signs, physical examination, and adverse events monitoring | Single-dose evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Christine Andersen, M.Sc., Study Director — Egalet A/S